CLINICAL TRIAL: NCT03369392
Title: The At-home Feasibility Evaluation of PANDA-Regional, a Smartphone Application Designed to Support Post-operative Pain Management in Patients Undergoing Peripheral Nerve Blocks
Brief Title: PANDA-Regional Feasibility Study of a Smartphone Pain Management Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Ron Ree, Clinical Associate Professor, University of British Columbia
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: H16-1196
Record Dates: First submitted 2017-11-28; First posted 2017-12-12 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Postoperative Pain; Anesthesia, Conduction
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Feasibility Cycle 1 (Experimental): Participants use the initial PANDA application.
  Interventions: Other: Panda application
- Feasibility Cycle 2 (Experimental): Participants use the PANDA application after modifications are made based on suggestions from participants in cycle 1.
  Interventions: Other: Panda application
- Feasibility Cycle 3 (Experimental): Participants use the PANDA application after modifications are made based on suggestions from participants in cycle 1 and 2.
  Interventions: Other: Panda application

INTERVENTIONS:
Other: Panda application — A smartphone-based postoperative pain management tool

SUMMARY:
Despite the numerous benefits of peripheral nerve blocks (PNBs) over general anesthesia (GA) in a variety of surgical procedures, PNBs can be associated with increased post-operative pain if pain medications are not taken correctly (titrated). Unfortunately, this is a common occurrence as patients often have difficulty titrating medications in the absence of direct medical care. PANDA, a smartphone-based postoperative pain management tool, is designed to address this issue by helping patients manage their pain medications. The purpose of this study is to demonstrate the feasibility of this application in patients who are discharged after receiving PNBs. The goal is to identify areas of improvement for the application itself. It is hypothesize that PANDA will be successful in supporting patients' postoperative pain management.

DETAILED DESCRIPTION:
As above

ELIGIBILITY:
Inclusion Criteria:

* Undergoing ambulatory surgical procedures that require peripheral nerve blocks for which there is an anticipated post-surgical pain model
* Planned post-discharge analgesic medications including non-steroidal anti-inflammatory drugs, acetaminophen and/or opioids for at least 2 days
* ASA I-III
* Written informed consent
* Have a smartphone device at their disposal

Exclusion Criteria:

* Inability or refusal to provide informed consent
* Presence of significant cognitive impairment, visual impairments, neurological injury, or psychomotor dysfunction that impairs ability to use the app
* Inability to follow study instructions and complete questionnaires in English

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of the PANDA application | 2-7 days post-operatively
  Measured by assessing the participants' compliance with the application in supporting ongoing pain assessments and analgesic administration.

SECONDARY OUTCOMES:
Identify usability issues | 2-7 days post-operatively
  Assessed by having participants complete a Computer Systems Usability Questionnaire (CSUQ) and a brief phone interview

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Ree, MD, Principal Investigator — University of British Columbia; Cynthia Fan, MD, Study Chair — University of British Columbia; Mark Ansermino, MBBCH, Study Chair — University of British Columbia; Terri Sun, MD, Study Chair — University of British Columbia; Lily Yu Long Chiu, MD, Study Chair — University of British Columbia; Dustin Dunsmuir, Study Chair — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dotto A, Dunsmuir D, Sun T, Chiu LYL, Ree R, Ansermino JM, Yarnold CH. The use of the Panda-Nerve Block pain app in single-shot peripheral nerve block patients: a feasibility study. Can J Anaesth. 2020 Sep;67(9):1140-1151. doi: 10.1007/s12630-020-01732-2. Epub 2020 Jun 4. PMID 32500515